CLINICAL TRIAL: NCT05467943
Title: A Multicenter, Open-label, Phase II Study to Evaluate the Efficacy, Safety and Pharmacokinetics of Tazemetostat for the Treatment of Patients With Relapsed/Refractory Follicular Lymphoma
Brief Title: Tazemetostat for the Treatment of Relapsed/Refractory Follicular Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hutchmed (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-TAZ-00CH1
Record Dates: First submitted 2022-06-28; First posted 2022-07-21 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Relapsed/Refractory Follicular Lymphoma With EZH2
MeSH Terms: conditions — Recurrence | interventions — tazemetostat

STUDY DESIGN:
Intervention Model Description: All patients will be enrolled to Cohort 1 and 2 based on the EZH2 mutations, respectively:
  * Cohort 1: MT patients with R/R FL; planned enrollment number: 19;
  * Cohort 2: WT patients with R/R FL; planned enrollment number: 20; Both cohorts have same dose administered: 800 mg, twice per day (BID), continuously, at a suggested interval of 12 hours between two doses.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohort 1 based on the EZH2 mutations (Experimental): MT patients with R/R FL; planned enrollment number: 19;
  Interventions: Drug: Tazemetostat
- Cohort 2 based on the EZH2 mutations, (Experimental): WT patients with R/R FL; planned enrollment number: 20;
  Interventions: Drug: Tazemetostat

INTERVENTIONS:
Drug: Tazemetostat — All patients will receive 800 mg of Tazemetostat, BID, administered in continuous 28-day therapeutic cycle

SUMMARY:
Treating Relapsed/Refractory Follicular Lymphoma with Tazemetostat

DETAILED DESCRIPTION:
This is an open-label, monotherapy, Phase II Study clinical study. The objective is to evaluate the efficacy, safety, and pharmacokinetics of Tazemetostat in the treatment of patients with relapsed/refractory follicular lymphoma. It is planned to enroll 39 Chinese patients in 2 cohorts.

ELIGIBILITY:
Inclusion Criteria:

1. Fully aware this study and signed the informed consent form in voluntary manner, and willing and able to comply with the study procedure;
2. Age ≥18 years;
3. Patients with histologically confirmed R/R FL (Grades 1, 2, 3a)
4. Patients must have one measurable lesion
5. Life expectancy ≥ 12 weeks;
6. Eastern Cooperative Oncology Group (ECOG) Performance Status 0 to 2
7. Adequate bone marrow function, renal function and hepatic function:
8. Currently human immunodeficiency virus (HIV), hepatitis B virus (HBV), hepatitis C virus (HCV) or cytomegalovirus (CMV) is inactive:
9. Female patients of childbearing potential must agree to adopt dual contraceptive method

Exclusion Criteria:

1. Previous use of Tazemetostat or other EZH2 inhibitors;
2. Patients with invasion of lymphoma to the central nervous system (CNS) or the pia mater;
3. Previous bone marrow malignancies,
4. Abnormalities associated with MDS and myeloproliferative neoplasms observed by cytogenetic testing and DNA sequencing;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2022-07-29 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
efficacy of Tazemetostat in EZH2 (MT) (Cohort 1) | 22 months
  Objective response rate (ORR) of Cohort 1 evaluated by the Independent Review Committee (IRC) [based on the International Working Group-Non-Hodgkin's Lymphoma [IWG-NHL] (Cheson) 2007]

SECONDARY OUTCOMES:
efficacy of Tazemetostat in EZH2 (WT) (Cohort 2) | 22 months
  Overall survival (OS) of Cohort 1 and 2. OS: defined as the time from the first dose of study drug to death for any cause.
safety of Tazemetostat in EZH2 (WT) (Cohort 2) | 22 months
  The incidence and severity of treatment emergent adverse events (TEAEs). Occurrence of AEs (including SAEs) will be monitored based on the changes in vital signs, physical examination, 12-lead ECG and laboratory examinations. The severity of AEs will be graded based on NCI CTCAE V5.0.
Geomean maximum concentration (Cmax) of tazemetostat and its metabolite EPZ-6930 in blood | Cycle1Day1: predose of first administration; 0.5, 1, 2, 4, 6, 8, and 12 hours postdose. Cycle1Day15: predose of first administration ; 0.5, 1, 2, 4, 6, 8, and 12 hours postdose. Cycle2Day1 and Cycle3Day1: predose of first administration.
  Cmax is defined as the maximum observed concentration that a drug achieves in a test area of the body after the drug has been administered. Plasma concentration-time profiles of tazemetostat and EPZ-6930 will be plotted using non-compartmental analysis and will be analyzed to determine Cmax. Cmax will be summarized as the geomean and geomean CV% for all participants.
Median time to reach maximum concentration (Tmax) of tazemetostat and its metabolite EPZ-6930 in blood | Cycle1Day 1: predose of first administration; 0.5, 1, 2, 4, 6, 8, and 12 hours postdose. Cycle1Day15: predose of first administration; 0.5, 1, 2, 4, 6, 8, and 12 hours postdose. Cycle2Day1 and Cycle3Day1: predose of first administration.
  Tmax is defined as the time from dosing to reach the maximum observed concentration a drug achieves in a specified compartment or test area of the body after the drug has been administered. Plasma concentration-time profiles of tazemetostat and EPZ-6930 will be plotted using non-compartmental analysis and will be analyzed to determine Tmax. Tmax will be summarized as the median (min, max) for all participants.
Geomean area under the drug concentration-time curve (AUC) of tazemetostat and its metabolite EPZ-6930 after administration of tazemetostat | Cycle1Day1: predose of first administration; 0.5, 1, 2, 4, 6, 8, and 12 hours postdose. Cycle1Day15: predose of first administration; 0.5, 1, 2, 4, 6, 8, and 12 hours postdose
  AUC represents the total drug exposure over a defined period of time. AUC will be calculated using the linear trapezoidal rule. Plasma concentrations of tazemetostat and EPZ-6930 will be analyzed using a non-compartmental analysis approach to determine individual participant estimates of AUC. AUC will be summarized as the geomean and geomean CV% for all participants.
Geomean minimum observed concentration at steady-state (Cmin) of tazemetostat and its metabolite EPZ-6930 in blood | Cycle1Day15, Cycle2Day1 and Cycle3Day1: predose of first administration
  Cmin is defined as the minimum observed concentration at steady-state during one dosing interval. Cmin will be summarized as the geomean and geomean CV% for all participants.

CONTACTS AND LOCATIONS:
Overall Officials: Junning Cao, MD, Principal Investigator — Shanghai Cancer Center
Locations (1):
- Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cao J, Chen G, Qiu L, Zhang L, Jiang M, Cheng Y, Zhang Q, Liu L, Li P, Shuang Y, Wang H, Xue H, Wu H, Zheng M, Zhou K, Li Z, Jing H, Yang W, Zhu Z, Li W, Wangwu J, Huang H, Jia Q, Chen D, Fan S, Shi MM, Su W. Efficacy and safety of tazemetostat, an EZH2 inhibitor, in Chinese patients with relapsed/refractory follicular lymphoma: a multicentre, single-arm, phase 2 study. EClinicalMedicine. 2025 Aug 18;87:103399. doi: 10.1016/j.eclinm.2025.103399. eCollection 2025 Sep. PMID 40896460